CLINICAL TRIAL: NCT05571124
Title: The Implementation of a Web-based Workplace Exercise Intervention in the Reduction of Spinal Pain in Sedentary Administrative Personnel: Protocol of a Mixed Methodology Study.
Brief Title: Workplace Exercise Intervention in Administrative Personnel to Reduce Spinal Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitat de Lleida (Other)
Responsible Party: Principal Investigator, Carlos Tersa Miralles, Tersa-Miralles C, Universitat de Lleida
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WEI
Record Dates: First submitted 2022-09-30; First posted 2022-10-07 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Back Pain; Sedentary Behavior
Keywords: Back Pain; Health Education; Therapeutic Exercise; Sedentary Behavior
MeSH Terms: conditions — Back Pain; Sedentary Behavior; Health Education

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: To ensure that allocation is concealed, one of the researchers will randomly create the codes in opaque envelopes with the username and password for participants to log into the web platform. The evaluators will be blinded to the data collection as each participant will be assigned a code for identification. The participants will not be blinded as they are aware of the intervention they are carrying out.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapeutic exercise (Experimental): It consists of implementing active breaks at the workstation through the use of the open source Learning Management System Sakai [33], It will be easy to use by the participants due to the platform is used by them in their daily work. Also, an administrative worker from the university will be involved in creating the modules where the content will be allocated to ensure that the navigation in the platform is user-friendly for them.musculoskeletal pathologies with sedentary lifestyles and maintained postures. The type of online application will depend on the results obtained in the qualitative phase, as we will adapt to the workers' preferences to facilitate accessibility to the content and make the experience as satisfactory as possible for them.
  Interventions: Behavioral: Therapeutic Exercise Intervention
- No intervention (No Intervention): Participants of the control group will be on a waiting list, encouraging them to maintain the same as usual in their daily activities and working hours. Once the intervention is finished, they will have access to the platform with the same content as the intervention group.

INTERVENTIONS:
Behavioral: Therapeutic Exercise Intervention — Participants will perform stretching and mobility exercises in short bouts of time.
  Other Names: Workplace exercise intervention; Active Breaks
  Arms: Therapeutic exercise

SUMMARY:
The goal of this Clinical trial is to compare treatments in sedentary administrative personnel with back pain. The main question it aims to answer:

The benefits of a workplace intervention with therapeutic exercise and pain education compared with only therapeutic exercise intervention

Participants will perform active pauses in their workplace with a web-based program that consists of videos or images of exercises and pain education information.

Researchers will compare a group Therapeutic exercise and pain education intervention with a group therapeutic exercise only to see if pain education plus exercise is a more beneficial intervention in reducing back pain in symptomatic administrative personnel.

DETAILED DESCRIPTION:
Introduction: Musculoskeletal pathologies are one of the leading causes of disability for the population worldwide, with office workers being one of the most affected groups. This study aims to design and implement a programme of therapeutic exercise and pain education in the workplace to reduce musculoskeletal pathology. The use of therapeutic exercise interventions at work is an economical and feasible option in which it is essential to consider biopsychosocial aspects when designing a successful treatment.

Methods: Mixed methodology study. Phase 1: A qualitative study with a phenomenological approach using semi-structured interviews to determine factors related to office workers' expectations about pain, maintaining static postures at work and implementing active breaks. Phase 2: Implementation of a Randomised Controlled Trial considering current scientific evidence and the results of the first phase with two intervention groups. A group in which therapeutic exercise will be performed at work with pain education, compared to a group implementing only exercise at the workplace.

Discussion: This study is a comprehensive and pragmatic intervention to implement therapeutic exercise in the workplace, considering workers' expectations regarding their pain and the implementation of active breaks. The use of digitalisation in the implementation of therapeutic exercise and pain education in office workers is a feasible and low-cost option. It can improve office workers' quality of life by increasing motivation and adherence to such interventions.

ELIGIBILITY:
Inclusion Criteria:

* More than 80% of the working day is in a seated position.
* Workers who have a computer or mobile device with an internet connection.
* Workers with more than three months of pain in the back area due to a non-specific cause.

Exclusion Criteria:-

* Part-time workers.
* Pathologies that cause chronic pain.
* Radiculopathies or symptomatic disc herniations/protrusions.
* Inability to perform low-moderate intensity exercise.
* People who are active in their daily lives outside of work willing to report that they meet the minimum stipulated by the WHO (a minimum of 10,000 steps per day and 75-150 minutes of vigorous-moderate physical activity per week).
* Undergoing physiotherapy treatment through public health or a private company.
* Workers on sick leave or during pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Reduction of Back Pain | Change from baseline back pain at six weeks
  The primary outcome to be analysed is back pain using the Visual Analogue Scale, a subjective assessment scale of intensity from 0 to 10, with 0 being "no pain" and 10 being "the worst possible pain".

SECONDARY OUTCOMES:
Back pain dysfunction | Change from baseline back pain dysfunction at six weeks
  Will be analysed using the Spanish version of the Spine Functional Index, a self-administered questionnaire in which the patient reports the state of his or her back concerning disability and dysfunction in daily activities.
Health related quality of life | Change from baseline quality of life at six weeks
  Will be analysed using the Spanish version of the EQ-5D-5L quality of life questionnaire which consists of 5 dimensions: mobility, self-care, activities of daily living, pain/discomfort and anxiety/depression.
Motivation of performing therapeutic exercise | Change from baseline motivation of performing therapeutic exercise at six weeks
  Motivation when performing the therapeutic exercise intervention will be analysed using the Spanish version of the questionnaire: Behavioural Regulation in Exercise Questionnaire-2.
Adherence to therapeutic exercise | Through study completion, an average of six weeks
  The percentage of open sessions and total video played of the participant will be analysed by the web analytics.

CONTACTS AND LOCATIONS:
Overall Officials: Esther Rubinat Arnaldo, PhD, Study Director — Universitat de Lleida; Francesc Rubi Carnacea, PhD, Study Director — Universitat de Lleida
Locations (1):
- Universitat de Lleida, Lleida, Catalonia, Spain

REFERENCES:
- [Background] GBD 2016 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 328 diseases and injuries for 195 countries, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet. 2017 Sep 16;390(10100):1211-1259. doi: 10.1016/S0140-6736(17)32154-2. PMID 28919117
- [Background] Sohrabi MS, Babamiri M. Effectiveness of an ergonomics training program on musculoskeletal disorders, job stress, quality of work-life and productivity in office workers: a quasi-randomized control trial study. Int J Occup Saf Ergon. 2022 Sep;28(3):1664-1671. doi: 10.1080/10803548.2021.1918930. Epub 2021 May 15. PMID 33870873
- [Background] Bevan S. Economic impact of musculoskeletal disorders (MSDs) on work in Europe. Best Pract Res Clin Rheumatol. 2015 Jun;29(3):356-73. doi: 10.1016/j.berh.2015.08.002. Epub 2015 Oct 24. PMID 26612235
- [Background] Koes BW, van Tulder MW, Thomas S. Diagnosis and treatment of low back pain. BMJ. 2006 Jun 17;332(7555):1430-4. doi: 10.1136/bmj.332.7555.1430. No abstract available. PMID 16777886
- [Background] Balague F, Mannion AF, Pellise F, Cedraschi C. Non-specific low back pain. Lancet. 2012 Feb 4;379(9814):482-91. doi: 10.1016/S0140-6736(11)60610-7. Epub 2011 Oct 6. PMID 21982256
- [Background] Janwantanakul P, Sihawong R, Sitthipornvorakul E, Paksaichol A. A Path Analysis of the Effects of Biopsychosocial Factors on the Onset of Nonspecific Low Back Pain in Office Workers. J Manipulative Physiol Ther. 2018 Jun;41(5):405-412. doi: 10.1016/j.jmpt.2017.10.012. Epub 2018 Jul 12. PMID 30007743
- [Background] Amiri S, Behnezhad S. Is job strain a risk factor for musculoskeletal pain? A systematic review and meta-analysis of 21 longitudinal studies. Public Health. 2020 Apr;181:158-167. doi: 10.1016/j.puhe.2019.11.023. Epub 2020 Feb 28. PMID 32059156
- [Background] Hoe VC, Urquhart DM, Kelsall HL, Zamri EN, Sim MR. Ergonomic interventions for preventing work-related musculoskeletal disorders of the upper limb and neck among office workers. Cochrane Database Syst Rev. 2018 Oct 23;10(10):CD008570. doi: 10.1002/14651858.CD008570.pub3. PMID 30350850
- [Background] Tersa-Miralles C, Bravo C, Bellon F, Pastells-Peiro R, Rubinat Arnaldo E, Rubi-Carnacea F. Effectiveness of workplace exercise interventions in the treatment of musculoskeletal disorders in office workers: a systematic review. BMJ Open. 2022 Jan 31;12(1):e054288. doi: 10.1136/bmjopen-2021-054288. PMID 35105632
- [Background] Luque-Suarez A, Martinez-Calderon J, Falla D. Role of kinesiophobia on pain, disability and quality of life in people suffering from chronic musculoskeletal pain: a systematic review. Br J Sports Med. 2019 May;53(9):554-559. doi: 10.1136/bjsports-2017-098673. Epub 2018 Apr 17. PMID 29666064
- [Background] Coggon D, Ntani G, Palmer KT, Felli VE, Harari R, Barrero LH, Felknor SA, Gimeno D, Cattrell A, Serra C, Bonzini M, Solidaki E, Merisalu E, Habib RR, Sadeghian F, Masood Kadir M, Warnakulasuriya SS, Matsudaira K, Nyantumbu B, Sim MR, Harcombe H, Cox K, Marziale MH, Sarquis LM, Harari F, Freire R, Harari N, Monroy MV, Quintana LA, Rojas M, Salazar Vega EJ, Harris EC, Vargas-Prada S, Martinez JM, Delclos G, Benavides FG, Carugno M, Ferrario MM, Pesatori AC, Chatzi L, Bitsios P, Kogevinas M, Oha K, Sirk T, Sadeghian A, Peiris-John RJ, Sathiakumar N, Wickremasinghe AR, Yoshimura N, Kelsall HL, Hoe VC, Urquhart DM, Derrett S, McBride D, Herbison P, Gray A. Disabling musculoskeletal pain in working populations: is it the job, the person, or the culture? Pain. 2013 Jun;154(6):856-63. doi: 10.1016/j.pain.2013.02.008. PMID 23688828
- [Background] Miles CL, Pincus T, Carnes D, Homer KE, Taylor SJ, Bremner SA, Rahman A, Underwood M. Can we identify how programmes aimed at promoting self-management in musculoskeletal pain work and who benefits? A systematic review of sub-group analysis within RCTs. Eur J Pain. 2011 Sep;15(8):775.e1-11. doi: 10.1016/j.ejpain.2011.01.016. Epub 2011 Feb 26. PMID 21354838
- [Background] Smith J, Faux SG, Gardner T, Hobbs MJ, James MA, Joubert AE, Kladnitski N, Newby JM, Schultz R, Shiner CT, Andrews G. Reboot Online: A Randomized Controlled Trial Comparing an Online Multidisciplinary Pain Management Program with Usual Care for Chronic Pain. Pain Med. 2019 Dec 1;20(12):2385-2396. doi: 10.1093/pm/pnz208. PMID 31498393
- [Background] Toelle TR, Utpadel-Fischler DA, Haas KK, Priebe JA. App-based multidisciplinary back pain treatment versus combined physiotherapy plus online education: a randomized controlled trial. NPJ Digit Med. 2019 May 3;2:34. doi: 10.1038/s41746-019-0109-x. eCollection 2019. PMID 31304380
- [Background] Palsson TS, Boudreau S, Hogh M, Herrero P, Bellosta-Lopez P, Domenech-Garcia V, Langella F, Gagni N, Christensen SW, Villumsen M. Education as a strategy for managing occupational-related musculoskeletal pain: a scoping review. BMJ Open. 2020 Feb 12;10(2):e032668. doi: 10.1136/bmjopen-2019-032668. PMID 32051307
- [Background] Devan H, Hale L, Hempel D, Saipe B, Perry MA. What Works and Does Not Work in a Self-Management Intervention for People With Chronic Pain? Qualitative Systematic Review and Meta-Synthesis. Phys Ther. 2018 May 1;98(5):381-397. doi: 10.1093/ptj/pzy029. PMID 29669089
- [Background] Louw A, Zimney K, Puentedura EJ, Diener I. The efficacy of pain neuroscience education on musculoskeletal pain: A systematic review of the literature. Physiother Theory Pract. 2016 Jul;32(5):332-55. doi: 10.1080/09593985.2016.1194646. Epub 2016 Jun 28. PMID 27351541
- [Background] Mills SEE, Nicolson KP, Smith BH. Chronic pain: a review of its epidemiology and associated factors in population-based studies. Br J Anaesth. 2019 Aug;123(2):e273-e283. doi: 10.1016/j.bja.2019.03.023. Epub 2019 May 10. PMID 31079836
- [Background] Slade SC, Patel S, Underwood M, Keating JL. What are patient beliefs and perceptions about exercise for nonspecific chronic low back pain? A systematic review of qualitative studies. Clin J Pain. 2014 Nov;30(11):995-1005. doi: 10.1097/AJP.0000000000000044. PMID 24300225
- [Background] Bull FC, Al-Ansari SS, Biddle S, Borodulin K, Buman MP, Cardon G, Carty C, Chaput JP, Chastin S, Chou R, Dempsey PC, DiPietro L, Ekelund U, Firth J, Friedenreich CM, Garcia L, Gichu M, Jago R, Katzmarzyk PT, Lambert E, Leitzmann M, Milton K, Ortega FB, Ranasinghe C, Stamatakis E, Tiedemann A, Troiano RP, van der Ploeg HP, Wari V, Willumsen JF. World Health Organization 2020 guidelines on physical activity and sedentary behaviour. Br J Sports Med. 2020 Dec;54(24):1451-1462. doi: 10.1136/bjsports-2020-102955. PMID 33239350
- [Background] O'Brien BC, Harris IB, Beckman TJ, Reed DA, Cook DA. Standards for reporting qualitative research: a synthesis of recommendations. Acad Med. 2014 Sep;89(9):1245-51. doi: 10.1097/ACM.0000000000000388. PMID 24979285
- [Background] Malterud K. Systematic text condensation: a strategy for qualitative analysis. Scand J Public Health. 2012 Dec;40(8):795-805. doi: 10.1177/1403494812465030. PMID 23221918
- [Background] Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S240-52. doi: 10.1002/acr.20543. No abstract available. PMID 22588748
- [Background] Cuesta-Vargas AI, Gabel CP. Validation of a Spanish version of the Spine Functional Index. Health Qual Life Outcomes. 2014 Jun 27;12:96. doi: 10.1186/1477-7525-12-96. PMID 24972525
- [Background] Hernandez G, Garin O, Pardo Y, Vilagut G, Pont A, Suarez M, Neira M, Rajmil L, Gorostiza I, Ramallo-Farina Y, Cabases J, Alonso J, Ferrer M. Validity of the EQ-5D-5L and reference norms for the Spanish population. Qual Life Res. 2018 Sep;27(9):2337-2348. doi: 10.1007/s11136-018-1877-5. Epub 2018 May 16. PMID 29767329
- [Background] Peugh JL, Strotman D, McGrady M, Rausch J, Kashikar-Zuck S. Beyond intent to treat (ITT): A complier average causal effect (CACE) estimation primer. J Sch Psychol. 2017 Feb;60:7-24. doi: 10.1016/j.jsp.2015.12.006. Epub 2016 Mar 24. PMID 28164801
- [Background] Jay K, Brandt M, Hansen K, Sundstrup E, Jakobsen MD, Schraefel MC, Sjogaard G, Andersen LL. Effect of Individually Tailored Biopsychosocial Workplace Interventions on Chronic Musculoskeletal Pain and Stress Among Laboratory Technicians: Randomized Controlled Trial. Pain Physician. 2015 Sep-Oct;18(5):459-71. PMID 26431123
- [Background] Hall G, Laddu DR, Phillips SA, Lavie CJ, Arena R. A tale of two pandemics: How will COVID-19 and global trends in physical inactivity and sedentary behavior affect one another? Prog Cardiovasc Dis. 2021 Jan-Feb;64:108-110. doi: 10.1016/j.pcad.2020.04.005. Epub 2020 Apr 8. No abstract available. PMID 32277997
- [Background] Kohl HW 3rd, Craig CL, Lambert EV, Inoue S, Alkandari JR, Leetongin G, Kahlmeier S; Lancet Physical Activity Series Working Group. The pandemic of physical inactivity: global action for public health. Lancet. 2012 Jul 21;380(9838):294-305. doi: 10.1016/S0140-6736(12)60898-8. PMID 22818941
- [Background] Powell KE, Paluch AE, Blair SN. Physical activity for health: What kind? How much? How intense? On top of what? Annu Rev Public Health. 2011;32:349-65. doi: 10.1146/annurev-publhealth-031210-101151. PMID 21128761
- [Background] Kirk MA, Rhodes RE. Occupation correlates of adults' participation in leisure-time physical activity: a systematic review. Am J Prev Med. 2011 Apr;40(4):476-85. doi: 10.1016/j.amepre.2010.12.015. PMID 21406284
- [Background] Edney S, Ryan JC, Olds T, Monroe C, Fraysse F, Vandelanotte C, Plotnikoff R, Curtis R, Maher C. User Engagement and Attrition in an App-Based Physical Activity Intervention: Secondary Analysis of a Randomized Controlled Trial. J Med Internet Res. 2019 Nov 27;21(11):e14645. doi: 10.2196/14645. PMID 31774402
- [Background] De Cocker K, Veldeman C, De Bacquer D, Braeckman L, Owen N, Cardon G, De Bourdeaudhuij I. Acceptability and feasibility of potential intervention strategies for influencing sedentary time at work: focus group interviews in executives and employees. Int J Behav Nutr Phys Act. 2015 Feb 18;12:22. doi: 10.1186/s12966-015-0177-5. PMID 25881297
- [Background] Gardner B, Smith L, Lorencatto F, Hamer M, Biddle SJ. How to reduce sitting time? A review of behaviour change strategies used in sedentary behaviour reduction interventions among adults. Health Psychol Rev. 2016;10(1):89-112. doi: 10.1080/17437199.2015.1082146. Epub 2015 Sep 16. PMID 26315814
- [Background] Ojo SO, Bailey DP, Hewson DJ, Chater AM. Perceived Barriers and Facilitators to Breaking Up Sitting Time among Desk-Based Office Workers: A Qualitative Investigation Using the TDF and COM-B. Int J Environ Res Public Health. 2019 Aug 14;16(16):2903. doi: 10.3390/ijerph16162903. PMID 31416112
- [Background] Ambrose KR, Golightly YM. Physical exercise as non-pharmacological treatment of chronic pain: Why and when. Best Pract Res Clin Rheumatol. 2015 Feb;29(1):120-30. doi: 10.1016/j.berh.2015.04.022. Epub 2015 May 23. PMID 26267006
- [Background] Booth J, Moseley GL, Schiltenwolf M, Cashin A, Davies M, Hubscher M. Exercise for chronic musculoskeletal pain: A biopsychosocial approach. Musculoskeletal Care. 2017 Dec;15(4):413-421. doi: 10.1002/msc.1191. Epub 2017 Mar 30. PMID 28371175
- [Background] Hadgraft NT, Brakenridge CL, LaMontagne AD, Fjeldsoe BS, Lynch BM, Dunstan DW, Owen N, Healy GN, Lawler SP. Feasibility and acceptability of reducing workplace sitting time: a qualitative study with Australian office workers. BMC Public Health. 2016 Sep 5;16(1):933. doi: 10.1186/s12889-016-3611-y. PMID 27595754
- [Background] de Wit M, Cooper C, Tugwell P, Bere N, Kirwan J, Conaghan PG, Roberts C, Aujoulat I, Al-Daghri N, Araujo de Carvalho I, Barker M, Bedlington N, Brandi ML, Bruyere O, Burlet N, Halbout P, Hiligsmann M, Jiwa F, Kanis JA, Laslop A, Lawrence W, Pinto D, Prieto Yerro C, Rabenda V, Rizzoli R, Scholte-Voshaar M, Vlaskovska M, Reginster JY. Practical guidance for engaging patients in health research, treatment guidelines and regulatory processes: results of an expert group meeting organized by the World Health Organization (WHO) and the European Society for Clinical and Economic Aspects of Osteoporosis, Osteoarthritis and Musculoskeletal Diseases (ESCEO). Aging Clin Exp Res. 2019 Jul;31(7):905-915. doi: 10.1007/s40520-019-01193-8. Epub 2019 Apr 16. PMID 30993659
- [Background] Biggs JS, Willcocks A, Burger M, Makeham MA. Digital health benefits evaluation frameworks: building the evidence to support Australia's National Digital Health Strategy. Med J Aust. 2019 Apr;210 Suppl 6:S9-S11. doi: 10.5694/mja2.50034. No abstract available. PMID 30927475
- [Background] Briggs AM, Cross MJ, Hoy DG, Sanchez-Riera L, Blyth FM, Woolf AD, March L. Musculoskeletal Health Conditions Represent a Global Threat to Healthy Aging: A Report for the 2015 World Health Organization World Report on Ageing and Health. Gerontologist. 2016 Apr;56 Suppl 2:S243-55. doi: 10.1093/geront/gnw002. PMID 26994264
- [Background] Rivilis I, Van Eerd D, Cullen K, Cole DC, Irvin E, Tyson J, Mahood Q. Effectiveness of participatory ergonomic interventions on health outcomes: a systematic review. Appl Ergon. 2008 May;39(3):342-58. doi: 10.1016/j.apergo.2007.08.006. Epub 2007 Nov 7. PMID 17988646
- [Derived] Tersa-Miralles C, Bravo C, Bellon F, Masbernat-Almenara M, Rubi-Carnacea F, Arnaldo ER. A web-based workplace exercise intervention among office workers with spinal pain: Protocol of a mixed methods study. PLoS One. 2025 Jun 9;20(6):e0325376. doi: 10.1371/journal.pone.0325376. eCollection 2025. PMID 40489458